CLINICAL TRIAL: NCT04733781
Title: Subcutaneous Injection of Large Volumes of Tumescent Lidocaine and Epinephrine (TLE) by Laypersons: a Double-blind, Non-inferiority, Randomized Clinical Trial
Brief Title: Subcutaneous Injection of Large Volumes of Tumescent Lidocaine and Epinephrine by Laypersons
Acronym: TLE-RCT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jeffrey Alan Klein, MD (Industry)
Responsible Party: Sponsor-Investigator, Jeffrey Alan Klein, MD, Principal Investigator, HK Surgical, Inc.
Organization: HK Surgical, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TLE-RCT
Record Dates: First submitted 2021-01-24; First posted 2021-02-02 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Venomous Snakebites; Local Anesthesia; Painless Injection; Regional Anesthesia; Dermatologic Surgery; Cutaneous Pain; Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Pain | interventions — Epinephrine

STUDY DESIGN:
Intervention Model Description: double-blind, non-inferiority, randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, Care Providers, Investigator and Outcome Assessors will not know the concentration of epinephrine, either 1mg/L or 2mg/L, in the tumescent solution of lidocaine (1gm/L) to be injected subcutaneous in a participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Subcutaneous injection of 125ml by a physician and self-injection of 125ml by a volunteer (Arm I): (Active Comparator): A volunteer layperson (research subject), at least 16 years of age, will first receive 125ml of TLE injected subcutaneously into the left anterior thigh by a physician. Then the subject will self-inject a second 125ml of TLE into his/her right anterior thigh.
  Interventions: Drug: Tumescent Lidocaine and Epinephrine
- Subcutaneous injection of 125ml by a physician and 125ml by another volunteer (Arm II): (Active Comparator): A volunteer layperson (primary research subject), at least 16 years of age, will first receive 125ml of TLE injected subcutaneously into the left anterior thigh by a physician. The primary research subject will then receive a second 125ml of TLE injected into his/her right anterior thigh by a second adult volunteer who is at least 16 years old and not a medical professional.
  Interventions: Drug: Tumescent Lidocaine and Epinephrine
- Subcutaneous injection of 250ml by a physician into a volunteer (Arm III) (Active Comparator): A volunteer layperson (research subject), at least 16 years old, will receive 250ml of TLE injected subcutaneously into the one anterior thigh by a physician.
  Interventions: Drug: Tumescent Lidocaine and Epinephrine

INTERVENTIONS:
Drug: Tumescent Lidocaine and Epinephrine — Subcutaneous injection of a relatively large volume (125ml to 250ml) of a relatively dilute solution of lidocaine (1gm/L) and epinephrine (1mg/L or 2mg/L).
  Other Names: Tumescent Local Anesthesia

SUMMARY:
This research is intended to show that it is safe and not difficult for nearly anyone to inject at least 125ml of a dilute solution of tumescent lidocaine and epinephrine (TLE), where a TLE solution consists of lidocaine (1gm/L) and epinephrine (1mg/L) in normal saline.

DETAILED DESCRIPTION:
The primary aim of this research is to demonstrate that of subcutaneous injection of tumescent (dilute) lidocaine and epinephrine (TLE) is safe, well tolerated, and easily performed by nearly anyone who is at least 16 years old. The primary aim will be achieved by conducting an IRB-approved double-blind, non-inferiority, randomized clinical trial (RCT).

The indications for TLE when injected into subcutaneous tissue are

* Pre-hospital treatment of a snakebite envenomation (SBE)
* Dermatologic surgical procedures totally by local anesthesia
* Pure sensory regional anesthesia for significant cutaneous and musculoskeletal pain.

The present TLE-RCT has three research Arms, which are as follows:

Injection of 125ml by a physician and self-injection of 125ml by a volunteer (Arm I): A volunteer layperson (research subject), at least 16 years of age, will first receive 125ml of TLE injected subcutaneously into the left anterior thigh by a physician. Then the subject will self-inject a second 125ml of TLE into his/her right anterior thigh.

Injection of 125ml by a physician and 125ml by another volunteer (Arm II): A volunteer layperson (primary research subject), at least 16 years of age, will first receive 125ml of TLE injected subcutaneously into the left anterior thigh by a physician. The primary research subject will then receive a second 125ml of TLE injected into his/her right anterior thigh by a second adult volunteer who is at least 16 years old and not a medical professional.

Injection of 250ml by a physician into a volunteer (Arm III) : A volunteer layperson (research subject), at least 16 years of age, will receive 250ml of TLE injected subcutaneously into the one anterior thigh by a physician.

There will be two TLE formulations, F1 and F2.

* F1 contains epinephrine 1mg/L = 1:1,000,000, or 0.25mg/250ml.
* F2 contains epinephrine 2mg/L = 1:500,000, or 0.5mg/250ml. F1 and F2 will both contain lidocaine 1gm/L = 0.1gm/100ml = 0.1% The maximum dose of dilute tumescent epinephrine in F1 and F2 is 0.25mg and 0.5mg, respectively. An EpiPen® contains 0.3mg of epinephrine. The concentration of epinephrine in an EpiPen® is 1:1000, which is 1000 and 500 times greater than the concentration of epinephrine in F1 and F2, respectively.

Individual subjects will be randomly assigned to receive either F1 or F2. The maximum dosage of tumescent lidocaine is 5mg/kg, which is clearly a safe dosage given that the risk of mild lidocaine toxicity at 28mg/kg of 0.1% TLE is 1 per 5,000,000

ELIGIBILITY:
Inclusion Criteria:

* All volunteer subjects will be healthy, mature in behavior and temperament, without mental impairment and at least 16 years of age.
* A volunteer TLE research subject must be a non-medical-professional layperson and must have signed an IRB-approved informed consent form prior to participation.
* All subjects must weigh at least 40kg = 88lb

Exclusion Criteria:

* Anyone who has a significant fear of needles or fear of injections
* A history of lidocaine allergy.
* A significant history of epinephrine hypersensitivity.
* History of an adverse reaction to percutaneous injections, such as fainting and lightheadedness (vasovagal reactions, near syncope).
* Significant needle phobia or anxiety.
* Vasovagal reaction associated with any medical procedures or the sight of blood.
* Uncontrolled or labile hypertension.
* Hyperthyroidism, thyroid medications.
* Recent phenylephrine (Actifed®) or pseudoephedrine use.
* Any significant cardiac arrhythmia including controlled atrial fibrillation tachycardia, mitral valve prolapse.
* Significant chronic renal impairment.
* Significant liver function abnormalities.
* History of having or having had a blood born infection with HIV, Hepatitis B, Hepatitis C.
* Evidence of active skin infection.
* Pregnant women are excluded.
* Subject has recently taken any drug(s) known to interfere with the metabolism of lidocaine such as erythromycin, clarithromycin, ketoconazole, fluconazole, sertraline (Zoloft), or ciprofloxacin.
* Subject has recently taken any drug known to interact adversely with epinephrine such as pseudoephedrine, ephedrine, or beta-blocker.
* History of radiation therapy or surgery involving the area near the proposed injection site.
* Pre-existing or concurrent infections (cutaneous, urinary, pneumonia are exclusionary).

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-02-22 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-07 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | up to 24 hours
  the incidence of any clinically significant adverse event associated with TLE injection, such as pain at injection site, vasovagal event, tachycardia, infection

SECONDARY OUTCOMES:
Numerical Pain Scale (NPS) | immediately after intervention
  Numerical Pain Scale (NPS) score following each injection, where the range of he scale is 0 to 10, and where 0= "no pain" and 10="worst imaginable pain"
Pulse Rate | up to 30 minutes after intervention
  Measure difference between pulse rates before and after subcutaneous injection of 250ml of TLE.
Blood Pressure Changes | up to 30 minutes after intervention
  Measure the differences between systolic and diastolic blood pressures before and after subcutaneous injection of 250ml of TLE.
EKG rhythm changes | up to 30 minutes after intervention
  EKG rhythm strips will be recorded before and after 250ml of TLE and any significant changes will be documented. Prior to the initial subcutaneous injection of the TLE solution, the EKG rhythm will be noted and recorded. For example, if the "pre-TLE" rhythm is "Normal Sinus Rhythm (NSR)" this observation will be recorded. After the subcutaneous TLE injection, a second EKG rhythm will be recorded. The analysis of the these two EKG rhythm strips will provide a dichotomous outcome variable: "no clinically significant EKG change" or "potentially significant EKG change." If there is a significant EKG rhythm strip change, then any relevant clinical details or observations will be recorded.
Human-Factors Associated with subcutaneous injection of a largfe volume of a TLE solution. | during the intervention
  Human-factor, or user interface difficulties encountered during the TLE injection process will be observed and a narrative of the observations will be recorded. The TLE-RCT is intended to demonstrate that any layperson can give a 125ml subcutaneous injection of a TLE in a manner that is safe and effective and essentially non-inferior to a similar injection administered by a physician. We will observe and record an apparent difficulties experience by the layperson when giving the injection. We will ask questions of the layperson to determine if the "instructions for use" are sufficient, and if not, we will record their suggestions for improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- HK Dermatology Care Center, San Juan Capistrano, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Other researcher, who wish to replicate our RCT-TLE trial will be provided with de-identified data upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available at the time that the data is first presented in a public forum.
Access Criteria: All information will be uploaded to www.tumescent.com
URL: http://www.tumescent.com

REFERENCES:
- [Background] Makdisi JR, Kim DP, Klein PA, Klein JA. Tumescent contravenom: murine model for prehospital treatment of Naja naja neurotoxic snake envenomation. Int J Dermatol. 2018 May;57(5):605-610. doi: 10.1111/ijd.13877. Epub 2018 Feb 20. PMID 29460967
- [Background] Klein JA, Jeske DR. Estimated Maximal Safe Dosages of Tumescent Lidocaine. Anesth Analg. 2016 May;122(5):1350-9. doi: 10.1213/ANE.0000000000001119. PMID 26895001
- [Background] Klein JA, Langman LJ. Prevention of Surgical Site Infections and Biofilms: Pharmacokinetics of Subcutaneous Cefazolin and Metronidazole in a Tumescent Lidocaine Solution. Plast Reconstr Surg Glob Open. 2017 May 30;5(5):e1351. doi: 10.1097/GOX.0000000000001351. eCollection 2017 May. PMID 28607871
- [Background] Klein JA. Tumescent technique for local anesthesia improves safety in large-volume liposuction. Plast Reconstr Surg. 1993 Nov;92(6):1085-98; discussion 1099-100. PMID 8234507
- [Background] Klein JA. The tumescent technique for liposuction surgery. J Am Acad Cosmetic Surg, 1987; 4:263-267.
- [Background] US Patent 10,786,483 B2. JA Klein, PA Klein, BA Klein. Tumescent Contravenom Drug Delivery (Sep 29, 2020).
- [Background] US Patent 10,493,024 B2. Klein. Tumescent infiltration drug delivery of high subcutaneous drug concentrations with prolonged local and systemic effects and minimal local or systemic toxicity (Dec 3, 2019).